CLINICAL TRIAL: NCT05412056
Title: A Randomized Double Blinded Controlled Trial of Using Metformin to Prevent Preterm Birth in Twin Pregnancy
Brief Title: Metformin to Prevent Preterm Birth in Twin Pregnancy
Acronym: TwinMet
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Mimi Seto, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UW 20-315
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Preterm Birth; Premature Obstetric Labor; Twin; Complicating Pregnancy; Pregnancy Complications; Pregnancy Preterm; Metformin; Drug Effect
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Pregnancy Complications | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Active Comparator): Metformin will be prescribed before 20 weeks to 33+6 weeks, started at a daily dose of 500mg in the first week, and the daily dose is increased by 500mg per week to a maximum of 2000mg in week 4 (1000mg twice per day). Women will be asked to take the maximum tolerated dose if they experience side effects from the medication.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo will be prescribed before 20 weeks to 33+6 weeks, started at a daily dose of 1 tablet in the first week, and the daily dose is increased by 1 tablet per week to a maximum of 4 tablets in week 4 (2 tablets twice per day). Women will be asked to take the maximum tolerated dose if they experience side effects from the medication.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin — as in arm/group description
  Arms: Metformin
Drug: Placebo oral tablet — as in arm/group description
  Arms: Placebo

SUMMARY:
Preterm birth (PTB) is a major challenge to perinatal health. It accounts for 75% of perinatal deaths and more than 50% of long-term neurological disabilities. Neonates born preterm are also at risk of significant comorbidities, for example respiratory distress syndrome, chronic lung disease, retinopathy of prematurity, necrotizing enterocolitis, intraventricular haemorrhage and sepsis in the short term, as well as cerebral palsy, motor and sensory impairment, learning difficulties, and increased risk of chronic disease in long run.

Twin pregnancy is associated with a higher risk of PTB when compared to singleton pregnancy. The National Vital Statistics reveals the PTB rate is 8.2% and 60.3% in singleton and twin pregnancy respectively in 2018. The mechanism of PTB in twin pregnancy is not completely understood and may be different from that of singleton pregnancy. At present, there are no good strategies to prevent PTB in twin pregnancy.

In singleton pregnancy, metformin has been used for the treatment of gestational diabetes in pregnant women with obesity/ overweight or polycystic ovarian syndrome (PCOS). The rate of PTB of pregnant women with PCOS is significantly lower after using metformin. A decreasing trend of PTB is also noted after metformin use in obese pregnant women without PCOS. There is no study to investigate the effect of metformin in twin pregnancy.

Premature uterine and amnion stretching in twin pregnancy can trigger preterm labour by increased prostaglandin synthesis and interleukin-1, activation of activator protein-1, expression of connexin-43 and stimulation of stretch dependent focal adhesion signaling. Inflammation is another risk factor for PTB. Metformin is an anti-inflammatory agent which can suppress inflammatory cytokines production and downregulate AMP-activated protein kinase medicated connexin-43 and nuclear factor κB activation. Anti-inflammatory actions of metformin can also reduce production of nitric oxide, prostaglandin E2 and pro-inflammatory cytokines through inhibition of NFκB activation in macrophages. Another possible mechanism to prevent PTB is the inhibition of mammalian target of rapamycin complex 1,which has a role in the timing of birth, by AMP-activated protein kinase. Therefore, metformin can be potentially used to prevent PTB in twin pregnancy. However, its effect in twin pregnancy has not been studied.

The objective of the study is to determine if the use of metformin in twin pregnancy can prevent PTB.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years old
* Viable twin pregnancy with dichorionic diamnioticity or monochorionic diamnioticity
* Gestational age less than 20 completed weeks

Exclusion Criteria:

* High order multiple pregnancy such as triplets or higher order multiple pregnancy with fetal reduction to twin pregnancy
* Monochorionic monoamniotic twin pregnancy
* Twin pregnancy with silent miscarriage of one twin
* Excessive vaginal bleeding
* Presence of congenital anomaly
* Rupture of membranes
* Congenital uterine anomaly
* Unwillingness or inability to comply with study procedures
* Known paternal or maternal abnormal karyotype
* Known renal, liver, or heart failure
* Pre-existing type 1 or 2 diabetes
* Treatment with metformin at the time of screening
* Allergic to metformin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | before 34+0 gestational weeks
  Number of participants with preterm birth

SECONDARY OUTCOMES:
Preterm birth | before 32+0 weeks
  Number of participants with preterm birth
Preterm birth | before 28+0 weeks
  Number of participants with preterm birth